CLINICAL TRIAL: NCT03032939
Title: The Effect of Tracheal Intubation Induced Autonomic Response on Photoplethysmography
Brief Title: The Effect of Tracheal Intubation on AC and DC Components of a Photoplethysmograph
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Pekka Talke, Professor of Anesthesia, University of California, San Francisco
Other Study IDs: PT071
Record Dates: First submitted 2017-01-24; First posted 2017-01-26 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: Anesthesia Intubation Complication
MeSH Terms: interventions — Intubation, Intratracheal

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: endotracheal intubation — standard endotracheal intubation of surgical patients after induction of anesthesia

SUMMARY:
Intraoperative stress responses (vasoconstriction and changes in heart rate) and postoperative pain can be monitored using photoplethysmography (PPG). PPG measures changes in tissue volume noninvasively. Therefore it can measure acute changes in arterial diameter (vasoconstriction). PPG signal has two components, AC and DC. Effects of noxious stimuli-induced stress responses (vasoconstriction) have not been studied on the DC component of PPG. The aim of this study was to investigate the effect of a known noxious stimulus (endotracheal intubation) on both the AC and DC components of PPG.

ELIGIBILITY:
Inclusion Criteria:

* Elective surgery
* General endotracheal anesthesia
* Over 18 years of age
* Healthy

Exclusion Criteria:

* Vascular disease
* Liver or kidney disease
* Overweight

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Elective, healthy surgical patients over 18 yrs of age
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2007-12-18 (Actual); Primary Completion 2012-01-30 (Actual); Study Completion 2015-01-30 (Actual)

PRIMARY OUTCOMES:
Photoplethysmography | within 60 seconds of intubation
  changes in AC and DC components of photoplethysmography

SECONDARY OUTCOMES:
Pulse rate | within 60 seconds of intubation
  Pulse rate from photoplethysmograph

CONTACTS AND LOCATIONS:
Overall Officials: Pekka O Talke, MD, Principal Investigator — University of California, San Francisco

IPD SHARING:
Plan to Share IPD: No
only a unique study number such as, IP01, that is unrelated to any patient identifiers will be used

REFERENCES:
- [Derived] Talke P. The Effect of Tracheal Intubation-Induced Autonomic Response on Photoplethysmography. Anesthesiol Res Pract. 2017;2017:7646541. doi: 10.1155/2017/7646541. Epub 2017 Apr 2. PMID 28469670